CLINICAL TRIAL: NCT05364567
Title: Vitamin D Supplementation in Patients With Vitiligo Induced Additive Effects With Phototherapy
Brief Title: Synergistic Effect of Vitamin D Supplementation in Patients With Vitiligo and Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Bo Young Chung, Principal Investigator, Clinical Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04-017
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Vitamin D Deficiency; Vitiligo
MeSH Terms: conditions — Vitamin D Deficiency; Vitiligo | interventions — Cholecalciferol; Phototherapy

STUDY DESIGN:
Intervention Model Description: All participants were randomly assigned to two groups: the control group and the study group. Both groups were treated with phototherapy including 308-nm excimer laser or narrowband ultraviolet B. Study group additionally had vitamin D supplementation through the injection of cholecalciferol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): They were treated with phototherapy including 308-nm excimer laser or narrowband ultraviolet B (NB-UVB). They had vitamin D supplementation through the injection of cholecalciferol additionally. The study group with vitamin D deficiency was treated with intramuscular injection of 200,000 IU cholecalciferol (Kwangdong Pharmaceutical Co., Seoul, Korea) once at baseline. Total study period was 6 months and the clinical assessments with checking adverse events were conducted every month.
  Interventions: Drug: cholecalciferol (vitamin D3); Procedure: Phototherapy
- Control group (Active Comparator): They were treated with phototherapy including 308-nm excimer laser or narrowband ultraviolet B (NB-UVB). Total study period was 6 months and the clinical assessments with checking adverse events were conducted every month.
  Interventions: Procedure: Phototherapy

INTERVENTIONS:
Drug: cholecalciferol (vitamin D3) — The study group with vitamin D deficiency was treated with intramuscular injection of 200,000 IU cholecalciferol (Kwangdong Pharmaceutical Co., Seoul, Korea) once at baseline.
  Arms: Study group
Procedure: Phototherapy — The phototherapy for treating depigmented areas was by using 308-nm xenon chloride excimer laser (E1, Jetema, Seoul, Korea) or NB-UVB (N-UVB 6000C, Choyang medical, Seongnam, Korea). The initial dose for excimer laser was decided based on the location of depigmented lesion with consideration of the previous results of the phototherapy;40-42 eye = 100mJ/cm2; head, face, ear, neck, axilla = 150mJ/cm2; arm, leg, trunk = 200mJ/cm2; wrist = 250mJ/cm2; elbow, knee = 300mJ/cm2; hand, foot = 400mJ/cm2; finger, toe = 600mJ/cm2; Meanwhile, initial dose for NB-UVB was 400mJ/cm2. If the erythema after laser disappears within 24 hours, the energy dose was increased by 50 mJ/cm2 for each treatment. But if the erythema sustained for 24-48 hours, the energy dose was maintained. If the erythema last longer than 48 hours, the energy dose was decreased by 50-100 mJ/cm2 at each session. If blistering or pain occured, the treatment was omitted until resolution of symptoms.

SUMMARY:
This prospective, randomized, controlled study was approved by the Institutional Review Board of Hallym University Kangnam Sacred Heart Hospital (IRB no. 2018-04-017). All study participants consented the study and agreed the written informed consent. All participants who are applicable to the inclusion criteria were randomly assigned to two groups: the control group and the study group. Both groups were treated with phototherapy including 308-nm excimer laser or narrowband ultraviolet B (NB-UVB). Study group had vitamin D supplementation through the injection additionally.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with non-segmental vitiligo based on clinical diagnosis.
2. patients who were ≥ 18 years old.
3. patients with lower serum vitamin D level (<20ng/mL).

Exclusion Criteria:

1. patients taking medicines such as thiazide, diuretics, lithium which can influence the serum vitamin D level.
2. pregnant or lactating women.
3. patients with diseases which can affect kidney such as chronic kidney disease, hyperparathyroidism, or hypoparathyroidism.
4. patients with uncontrolled chronic diseases like diabetes mellitus, hyperlipidemia, hypertension
5. patients whose spot urine calcium level was over 30mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Vitiligo Area Scoring Index (VASI) | baseline
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 1 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 2 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 3 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 4 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 5 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.
Vitiligo Area Scoring Index (VASI) | 6 month
  Each VASI score was decided by multiplying the area of vitiligo and the extent of depigmentation.

SECONDARY OUTCOMES:
Physician global assessment (PGA) | baseline
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 1 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 2 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 3 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 4 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 5 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.
Physician global assessment (PGA) | 6 month
  The PGA score was calculated to check the improvement after treatments. The scale was evaluated on a scale from 0 to 4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = 76-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Chung, M.D., PhD, Study Chair — Department of Dermatology, Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No